CLINICAL TRIAL: NCT05631002
Title: Chemical Shift Encoding-based Water-fat Magnetic Resonance Imaging in Spinal Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022403
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-08

CONDITIONS: Spinal Tumor; Bone Tumor
MeSH Terms: conditions — Spinal Cord Neoplasms; Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with benign spinal tumor
  Interventions: Diagnostic Test: Chemical shift encoding-based water-fat MRI
- Patients with intermediate spinal tumor
  Interventions: Diagnostic Test: Chemical shift encoding-based water-fat MRI
- Patients with malignant spinal tumor
  Interventions: Diagnostic Test: Chemical shift encoding-based water-fat MRI

INTERVENTIONS:
Diagnostic Test: Chemical shift encoding-based water-fat MRI — Chemical shift encoding-based water-fat magnetic resonance imaging (MRI): a non-invasive method

SUMMARY:
Fat composition of the spinal tumors is positively correlated with classification and differential diagnosis of benign and malignant tumors.

DETAILED DESCRIPTION:
Chemical shift encoding-based water-fat magnetic resonance imaging (MRI) is a non-invasive method that provides quantitative information about the biochemical water-fat composition of bone marrow and skeletal muscle in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Pathological biopsy of a patient with diagnosed spinal tumor lesion, and preoperative examination Chemical shift encoding-based water-fat MRI was performed.

Exclusion Criteria:

* Recurrent neoplasms; Lesion diameter < 1 cm; Poor image quality.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with spinal tumors
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Type of tumor | One month before treatment
  Pathological diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Ning Lang, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided